CLINICAL TRIAL: NCT05281107
Title: Vitamin D Supplementation, Parathyroid Hormone (PTH) and Plasma Vitamin D Response Among Malaysian Female Adults: Double Blinded, Randomised Clinical Trial of Efficacy
Brief Title: Vitamin D Supplementation and PTH Response Among Malaysian Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Melissa Leong En Ying, Principal Investigator, IMU University, Malaysia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: IMU R 144/2014 - File II
Record Dates: First submitted 2022-02-28; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo, 500 mg calcium (Placebo Comparator): Participants received 500 mg calcium in berry flavoured sachet powder daily for 16 weeks
  Interventions: Dietary Supplement: Placebo, 500 mg calcium; Dietary Supplement: 600 IU vitamin D + 500 mg calcium; Dietary Supplement: 1200 IU vitamin D + 500 mg calcium; Dietary Supplement: 4000 IU vitamin D + 500 mg calcium
- 600 IU vitamin D + 500 mg calcium (Active Comparator): Participants received 600 IU vitamin D with 500 mg calcium in berry flavoured sachet powder daily for 16 weeks
  Interventions: Dietary Supplement: Placebo, 500 mg calcium; Dietary Supplement: 600 IU vitamin D + 500 mg calcium; Dietary Supplement: 1200 IU vitamin D + 500 mg calcium; Dietary Supplement: 4000 IU vitamin D + 500 mg calcium
- 1200 IU vitamin D + 500 mg calcium (Active Comparator): Participants received 1200 IU vitamin D with 500 mg calcium in berry flavoured sachet powder daily for 16 weeks
  Interventions: Dietary Supplement: Placebo, 500 mg calcium; Dietary Supplement: 600 IU vitamin D + 500 mg calcium; Dietary Supplement: 1200 IU vitamin D + 500 mg calcium; Dietary Supplement: 4000 IU vitamin D + 500 mg calcium
- 4000 IU vitamin D + 500 mg calcium (Active Comparator): Participants received 4000 IU vitamin D with 500 mg calcium in berry flavoured sachet powder daily for 16 weeks
  Interventions: Dietary Supplement: Placebo, 500 mg calcium; Dietary Supplement: 600 IU vitamin D + 500 mg calcium; Dietary Supplement: 1200 IU vitamin D + 500 mg calcium; Dietary Supplement: 4000 IU vitamin D + 500 mg calcium

INTERVENTIONS:
Dietary Supplement: Placebo, 500 mg calcium — Berry flavoured sachet powder (500 mg calcium)
Dietary Supplement: 600 IU vitamin D + 500 mg calcium — Berry flavoured sachet powder (600 IU vitamin D + 500 mg calcium)
Dietary Supplement: 1200 IU vitamin D + 500 mg calcium — Berry flavoured sachet powder (1200 IU vitamin D + 500 mg calcium)
Dietary Supplement: 4000 IU vitamin D + 500 mg calcium — Berry flavoured sachet powder (4000 IU vitamin D + 500 mg calcium)

SUMMARY:
This clinical trial was designed to determine the efficacy of vitamin D supplementation on plasma 25-hydroxyvitamin D [25(OH)D] and intact parathyroid hormone (PTH) concentrations of Malaysian female adults of child-bearing age after daily intake of vitamin D supplements containing either 0 IU, 600 IU, 1200 IU or 4000 IU vitamin D for 16 weeks.

DETAILED DESCRIPTION:
After being informed regarding the study protocol and requirements, participants given informed consent were interviewed using a questionnaire for collection of background data and medical history as a screening process. Eligible participants were randomly assigned in a double-blind manner to receive daily 500 mg of calcium with either 0, 600 IU, 1200 IU or 4000 IU vitamin D supplement for 16 weeks. Questionnaires and anthropometric measurements were collected at baseline and post 16 weeks supplementation trial. Primary outcomes of plasma 25(OH)D and intact PTH were measured via fasting intravenous blood samples at baseline and post 16 weeks trial.

ELIGIBILITY:
Inclusion Criteria:

* three major ethnic groups (Malay, Chinese, Indian)
* age 20-45 years

Exclusion Criteria:

* any diseases or conditions that may affect vitamin D metabolism, such as diabetes, cardiovascular diseases, bone diseases, autoimmune diseases, had major gastrointestinal surgery and diagnosed primary hyperparathyroidism
* medications that might affect vitamin D metabolism, such as insulin, thiazide diuretics, prednisolone, biphosphonates, tamoxifen and phenytoin
* pregnant and lactating women

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasma 25-hydroxyvitamin D at week 16 | Baseline and week 16
  5ml of fasting blood sample were taken by venepuncture into heparin tubes. Collected blood samples were centrifuged at 4000 rpm for 10 minutes, extracted plasma and stored at -80˚C until sent for analysis

SECONDARY OUTCOMES:
Change from baseline intact parathyroid hormone at week 16 | Baseline and week 16
  5ml of fasting blood sample were taken by venepuncture into heparin tubes. Collected blood samples were centrifuged at 4000 rpm for 10 minutes, extracted plasma and stored at -80˚C until sent for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Geok Lin Khor, Study Chair — IMU University, Malaysia; Megan Chong, Study Director — IMU University, Malaysia
Locations (1):
- International Medical University, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because of shared IPs. Data are available from the International Medical University Institutional Data Access (contact via khor.geoklin@gmail.com) for researchers who meet the criteria for access to confidential data

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT05281107/Prot_SAP_ICF_000.pdf